CLINICAL TRIAL: NCT04513509
Title: The Surrogate Marker of Rate Control in Patients With Atrial Fibrillation
Brief Title: Rate Control in Patients With Atrial Fibrillation
Acronym: RaP-AF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 202006205RIND
Record Dates: First submitted 2020-08-09; First posted 2020-08-14 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Atrial Fibrillation; Rate Control; Cardiopulmonary Exercise Test
Keywords: Atrial Fibrillation; rate control; cardiopulmonary exercise test
MeSH Terms: conditions — Atrial Fibrillation | interventions — Atenolol; Bisoprolol; Metoprolol; Nebivolol; Propranolol; Diltiazem; Verapamil; Digoxin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- rate control (Experimental)
  Interventions: Drug: Atenolol, Bisoprolol, Metoprolol, Nebivolol, Propranolol, Diltiazem, Verapamil, digoxin

INTERVENTIONS:
Drug: Atenolol, Bisoprolol, Metoprolol, Nebivolol, Propranolol, Diltiazem, Verapamil, digoxin — Start with empirical lower dose for 3 months, and then titrate up

SUMMARY:
To search for the best marker for the patients in atrial fibrillation with rate control

DETAILED DESCRIPTION:
In an aging society, the prevalence of atrial fibrillation is increasing. The main treatment strategy is to reduce the complications of embolic stroke and heart failure. Among these patients, a group of them will choose to have "rate control" based on the heart conditions and the preference of the patients. The strategy is to control the ventricular rate by drugs to prevent the heart from failure. However, when the physicians attempt to do so, they encounter two questions: how much is the optimal drug dose? And what is the best marker we are looking to? To answer these questions, the investigators design a prospective, cross-over study to explore this issue. The participants will do cardiopulmonary exercise test (CPET) before and after treatment. They will receive another CPET if drug dose is titrated up. With the study, the investigators will understand whether a resting heart rate can be a good marker for optimal drug dosage, and what is the optimal range of heart rate the physicians should target.

ELIGIBILITY:
Inclusion Criteria:

1. 18~90 years old
2. Rate control is preferred after shared decision making

Exclusion Criteria:

1. cannot cooperate with or complete CPET
2. has contraindication for CPET, such as uncontrolled heart failure, hypertension, angina, valvular heart disease, lung function impariment that SaO2<90% at room air.
3. Ventricular rate below 80/min before any medication
4. Permanent pacemaker implanted

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2020-10-21 (Actual); Primary Completion 2022-06-21 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Change of Maximal Oxygen consumption | 0, 3, 6 months
  acquire the data by Cardiopulmonary exercise test (CPET) with different (low and high) drug dosages for rate control

CONTACTS AND LOCATIONS:
Overall Officials: Chih-Chieh Yu, MD.PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan